CLINICAL TRIAL: NCT05769387
Title: Multihormonal Deficiencies and miRNA Profile in Chronic Heart Failure: Effects of Combined Hormonal Replacement Therapy
Status: Completed | Type: Observational
Sponsor: IRCCS SYNLAB SDN (Other)
Responsible Party: Sponsor
Other Study IDs: 5-18
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Patients With Ischemic or Idiopathic Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with no hormonal deficit
- Patients with hormonal deficiencies

SUMMARY:
The results from this study will be useful to gain detailed information on the correlation related to pathophysiological aspects between endocrine system and clinical status of patients with heart failure, and to identify factors correlated with the progression and prognosis of ICC

ELIGIBILITY:
Inclusion Criteria:

* ischemic or idiopathic dilated cardiomyopathy, stable medications for at least three months including ß-blocker that must be started at least 6 months before entering the study, fraction of left ventricular ejection less than or equal to 49%

Exclusion Criteria:

* Age < 18 years, Inability to perform a bicycle ergometer exercise test. Diabetes mellitus in poor glycometabolic control and/or proliferative retinopathy or nonproliferative retinopathy severe grade. Severe renal failure; Hepatic cirrhosis advanced. Active neoplastic disease or history of malignancy. Patients with severe acute illness caused by complications from open heart or abdominal surgery, multiple accidental trauma, or acute respiratory failure. Active infection or sepsis. Any allergies to growth hormone, testosterone, vitamin D, or other excipients such as benzyl alcohol, sucrose, phosphoric acid, sodium hydroxide, or methacresol. Acute Coronary Syndrome within the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Enrollment of no. 250 subjects with CCI. The patients will be recruited from among patients belonging to the UOC of Internal Medicine with Cardiology and Respiratory Address of the AOU Federico II in Naples and the Division of Cardiology "San Giovanni di Dio and Ruggi d'Aragona" Salerno
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2022-05-22 (Actual)

PRIMARY OUTCOMES:
Evaluation of the association between hormonal deficits (single or multiple), miRNA profile and clinical/functional indices in patients with heart failure | 1-48 months
  Patients will be followed with the goal of determining whether the deficits hormonal deficits have an impact on prognosis. In the pilot study, a significant benefit is expected in terms of improved quality of life and physical performance of patients following adequate hormone replacement treatment. In addition, the clinical relevance of the association between anabolic deficits (single or multiple), miRNA expression profile, vitamin D levels, and clinical/functional indices in patients with HCI in order to identify novel biomarkers for the progression of human collagenase inhibitor HCI
Evaluation of clinical and morphological effects where necessary in patients With multiple hormonal deficits in addition to standard medical therapy | 1-48 months
  Evaluation of the prognostic impact of hormone deficits and miRNA levels in a large population of heart failure patients

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Synlab SDN, Naples, Italy